CLINICAL TRIAL: NCT05309486
Title: Effects of Online Pilates and Face-To-Face Pilates on Healthy Individuals During the COVID-19 Pandemic: A Randomized Controlled Study
Brief Title: Effects of Online Pilates and Face-To-Face Pilates on Healthy Individuals
Acronym: COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Bulguroglu, Assistant Professor, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Healthy Lifestyle; Health Behavior
Keywords: Online pilates; Quality of life; Depression; Core; Pilates exercises
MeSH Terms: conditions — Health Behavior; Depression

STUDY DESIGN:
Intervention Model Description: Using a computer program, the investigators randomly placed individuals who completed the initial assessment into the online pilates group (OPG) or face-to-face pilates group (FPG).
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were evaluated at the beginning of the study and 8 weeks later by an experienced physical therapist blind to randomization. The group participants belonged to was not disclosed to the participants from the initial assessment to the end.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online pilates group (Experimental): Online pilates, which lasts for eight weeks, three days a week for 1 hour, will be carried out by Australian Pilates and Physiotherapy Institute certified and experienced Ph.D. Physiotherapist Halil Ibrahim Bulguroglu. Microsoft Teams program will be used to implement the online practice method. The individuals in both pilates exercise groups will be divided into six small groups of 3 or 4 people to make the exercises more effective. In this study, the program will be 15 minutes of warm-up, 30 minutes of pilates, and 15 minutes of cool-down and stretching exercises. The exercises will be performed in ten repetitions. The same exercises will be applied in online pilates and face-to-face pilates trainings.
  Interventions: Other: Online and Face-to-face Pilates trainings
- Face-to-face pilates group (Active Comparator): Face-to-face pilates training, which lasts for a total of 8 weeks, 3 days a week for 1 hour, will be carried out by Australian Pilates and Physiotherapy Institute certified and experienced Ph.D. Physiotherapist Halil Ibrahim Bulguroglu. Face-to-face pilates training will be held at Ankara Medipol University. To make the exercises more effective, the individuals in both pilates exercise groups will be divided into six small groups of 3 or 4 people. In this study, the program will be 15 minutes of warm-up, 30 minutes of pilates exercises, 15 minutes of cool-down and stretching exercises, and the exercises will be performed as 10 repetitions. The same exercises will be applied in online pilates and face-to-face pilates trainings.
  Interventions: Other: Online and Face-to-face Pilates trainings

INTERVENTIONS:
Other: Online and Face-to-face Pilates trainings — Key elements of Pilates, including breathing, focusing, rib cage position, shoulder position, and head and neck positions, will be taught in both groups on the first day. Individuals will be asked to maintain the smoothness of these critical elements throughout the exercises. Different imagery techniques will be used in the exercises, and the exercises will be combined with breathing exercises. The intensity of the exercises will be increased by using different positions and elastic bands (Theraband Elastic Band Hygienic Corporation, Akron, Ohio). Band Resistances will be increased in biweekly periods. Stretching and posture exercises will be used during the cool-down period. The subjects in pilates group will be informed about the side effects such as shortness of breath, dizziness, headache, and muscle pain. Participants will be asked to stop the exercise in case of any side effects.

SUMMARY:
Many studies on pilates have shown that these exercises positively affect the endurance of core muscles, mental health, and quality of life in healthy individuals when applied face-to-face.

In a few recent studies, the effects of online pilates training have been examined and shown to be effective on core endurance, depression, and quality of life. In the results of these studies, it has been emphasized that it is necessary to compare whether online pilates training is as practical as face-to-face pilates training. For this reason, the investigators thought that randomized controlled studies investigating the effects of online and face-to-face pilates methods in healthy individuals are needed. The investigators planned a randomized controlled study investigating the impact of online pilates and face-to-face pilates methods. The study aims to examine and compare the effects of online pilates and face-to-face pilates methods on core muscle endurance, depression, and quality of life in healthy individuals.

DETAILED DESCRIPTION:
An experienced physiotherapist blind will evaluate participants by randomization at the start of the study and eight weeks later. The group participants belong to will not be disclosed to the participants until the end of the first assessment. Individuals who complete the initial evaluation will be randomly assigned to the online pilates group (OPG) or face-to-face pilates group (FPG) using a computer program. Both online and face-to-face applications will be carried out under the supervision of a physiotherapist with 11 years of experience.

Participants included in the study will be evaluated with data collection forms filled twice, before and after the training programs. The participants' demographic information (age, body weight, height, body mass index) will be recorded.

Statistical analysis will be performed using SPSS software, version 21 (SPSS Inc. Chicago, IL, USA). The normal distribution of the variables will be determined using histograms, probability plots, and the Shapiro-Wilk test. Due to the abnormal distribution, the median and interquartile range (IQR) will be used for descriptive statistics. A Mann-Whitney U test will be used to compare baseline and vary values between groups. The Wilcoxon test will compare baseline values within the group to values after six weeks. The significance level will be set-top < 0.05 for all analyses. Effect sizes will be evaluated according to Cohen's d standards within pre-post differences. Effect size results will be interpreted as small (≥ 0.2), moderate (≥ 0.5), or large (≥ 0.8) according to the guidelines.

ELIGIBILITY:
Inclusion Criteria:

* 25-40 years of age.
* Voluntarily participate in research to accept

Exclusion Criteria:

* Any cardiovascular, orthopedic, visual, hearing, and perception problems that may affect the results of the research.
* Participating in other exercises or physiotherapy programs during the past 6 months.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-05-21 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Core muscle endurance- Baseline | Assessment will be conducted before the intervention
  Mcgill core endurance tests
Core muscle endurance- Post intervention | Assessment will be conducted immediately after the intervention
  Mcgill core endurance tests
Depression - Baseline | Assessment will be conducted before the intervention
  Beck Depression Scale (BDI). The score range in BDI, which is a 21-item self-evaluation type scale, is 0-63.
Depression - Post intervention | Assessment will be conducted immediately after the intervention
  Beck Depression Scale (BDI). The score range in BDI, which is a 21-item self-evaluation type scale, is 0-63.
Quality of life - Baseline | Assessment will be conducted before the intervention
  Short Form-36 (SF-36). SF-36; consists of 36 items to measure eight dimensions such as physical, mental, and general health. In the subscales evaluated between 0 and 100, a high score indicates a good quality of life.
Quality of life - Post intervention | Assessment will be conducted immediately after the intervention
  Short Form-36 (SF-36). SF-36; consists of 36 items to measure eight dimensions such as physical, mental, and general health. In the subscales evaluated between 0 and 100, a high score indicates a good quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: HALIL IB BULGUROGLU, PHD PT, Principal Investigator — Ankara Medipol University
Locations (1):
- Ankara Medipol University, Altındağ, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Quiles-Sanchez LV, Baroutas I, Kyriakos G, Gravvanis N, Georgakopoulou VE, Trakas N, Damaskos C, Garmpi A, Garmpis N, Antoniou V, Farmaki P, Patsouras A, Voutyritsa E, Diamantis E. Medical Flossing and the Pilates Method: Their Effectiveness on the Strength, Endurance, and Functionality of Healthy Individuals. Cureus. 2021 Apr 29;13(4):e14758. doi: 10.7759/cureus.14758. PMID 34084682
- [Result] Lemos AQ, Brasil CA, Valverde D, Ferreira JDS, Lordelo P, Sa KN. The pilates method in the function of pelvic floor muscles: Systematic review and meta-analysis. J Bodyw Mov Ther. 2019 Apr;23(2):270-277. doi: 10.1016/j.jbmt.2018.07.002. Epub 2018 Jul 10. PMID 31103107
- [Result] Rimmer JH, Thirumalai M, Young HJ, Pekmezi D, Tracy T, Riser E, Mehta T. Rationale and design of the tele-exercise and multiple sclerosis (TEAMS) study: A comparative effectiveness trial between a clinic- and home-based telerehabilitation intervention for adults with multiple sclerosis (MS) living in the deep south. Contemp Clin Trials. 2018 Aug;71:186-193. doi: 10.1016/j.cct.2018.05.016. Epub 2018 May 30. PMID 29859267
- [Result] Suner-Keklik S, Numanoglu-Akbas A, Cobanoglu G, Kafa N, Guzel NA. An online pilates exercise program is effective on proprioception and core muscle endurance in a randomized controlled trial. Ir J Med Sci. 2022 Oct;191(5):2133-2139. doi: 10.1007/s11845-021-02840-8. Epub 2021 Oct 30. PMID 34716884
- [Result] Campos RR, Dias JM, Pereira LM, Obara K, Barreto MS, Silva MF, Mazuquin BF, Christofaro DG, Fernandes RA, Iversen MD, Cardoso JR. Effect of the Pilates method on physical conditioning of healthy subjects: a systematic review and meta-analysis. J Sports Med Phys Fitness. 2016 Jul-Aug;56(7-8):864-73. Epub 2015 May 25. PMID 26004043
- [Result] Cruz-Ferreira A, Fernandes J, Laranjo L, Bernardo LM, Silva A. A systematic review of the effects of pilates method of exercise in healthy people. Arch Phys Med Rehabil. 2011 Dec;92(12):2071-81. doi: 10.1016/j.apmr.2011.06.018. Epub 2011 Oct 24. PMID 22030232
- [Derived] Bulguroglu HI, Bulguroglu M. The effects of online pilates and face-to-face pilates in healthy individuals during the COVID-19 pandemic: a randomized controlled study. BMC Sports Sci Med Rehabil. 2023 Feb 2;15(1):12. doi: 10.1186/s13102-023-00625-3. PMID 36732823